CLINICAL TRIAL: NCT02956291
Title: Multi-Parametric Quantitative MR Imaging in Evaluation of Brain Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE8316
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor
Keywords: glioma; brain tumor; brain metastasis
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Newly Diagnosed Brain Tumors (Experimental): Participants with newly diagnosed brain tumors will undergo Magnetic Resonance Fingerprinting (MRF) scan along with their clinical scan, followed by standard of care surgery, radiation, and chemotherapy. Follow-up MRF scans will be performed to visualize recurrence.
  Interventions: Device: Magnetic Resonance Fingerprinting
- Treated tumors with possible recurrence (Experimental): Participants with treated brain tumors with possible recurrence will undergo Magnetic Resonance Fingerprinting (MRF) scan along with their clinical scan, followed by standard of care surgery, radiation, and chemotherapy. Follow-up MRF scans will be added to the repeat MRI studies as determined appropriate by the referring physician/primary care team.
  Interventions: Device: Magnetic Resonance Fingerprinting

INTERVENTIONS:
Device: Magnetic Resonance Fingerprinting — Non-contrast MRF acquisition will be acquired through the region of tumor in all patients. For patients receiving intravenous gadolinium based contrast, a post contrast MRF acquisition will also be acquired. This acquisition will be skipped in patients who do not receive or are not eligible for receiving IV contrast as a part of their clinical scan. The research scan will take approximately 10-15 minutes
  Other Names: MRF; 3D-MRF; MRF relaxometry

SUMMARY:
The purpose of the research study is to test new methods that could improve diagnosis and assessment of brain tumors. One of these methods is a new MR (magnetic resonance) imaging technique called magnetic resonance fingerprinting (MRF), which allows for rapidly scanning the patient and provides quantitative information on tumor tissue. The investigators will compare the data gathered from MR Fingerprinting with other imaging tests, clinical information, treatment details and biopsy results to evaluate the accuracy of this new technique.

DETAILED DESCRIPTION:
The primary objective of this study is to 1) evaluate the utility of quantitative MRI imaging including 3D-MRF in differentiating among different brain tumors and differentiating recurrent brain tumor (TR) from treatment effects

Secondary objectives include evaluating the correlation between quantitative MRI imaging with histopathological characteristics and genetic markers in pre-therapy setting and with treatment response and clinical outcomes in post treatment setting.

GROUP 1: All patients with newly diagnosed intra-axial brain neoplasms undergo volumetric MRI study with contrast for surgical planning or clinical diagnosis. Diffusion, diffusion tensor imaging and perfusion imaging are often performed as a part of standard clinical imaging. In addition to these acquisitions, the research 3D-MRF acquisition through the entire tumor will be acquired. The imaging parameters will be correlated individually and in combination with biopsy/ resection outcomes.

GROUP 2: All patients with brain tumors who present at post therapy follow up with imaging progression undergo serial imaging as a part of clinical care. The research 3D-MRF acquisitions will be added to these clinical scans. All the quantitative parameters will be evaluated individually and in combination to differentiate post treatment changes from tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intra-axial brain tumor at initial diagnosis or patients with known treated brain tumors on follow-up with concern for imaging progression
* Ability to understand and the willingness to sign a written informed consent document, or, in cases where the patient may have cognitive impairment, consent by a legal authorized representative or power of attorney
* Patients with brain metastases undergoing partial brain radiation (gamma knife or SRS) with ability to undergo research scan at baseline, 1 month and , 3 months, and 6 months

Exclusion Criteria:

* Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips.
* The presence of an implanted pacemaker or implanted defibrillator device.
* Patients with contraindications for MRI due to embedded foreign metallic objects. Bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient.
* Pregnancy. Regular clinical practice already excludes pregnant patients from gadolinium contrast.
* Implanted medical device not described above that is not MRI-compatible.
* Known history of severe claustrophobia.
* Prisoners and members of other vulnerable populations will be excluded from this study. The subject selection population will not regularly include prisoners and other vulnerable population members as these populations will not provide any additional unique information to or uniquely benefit from the study. Non-English speaking population will be excluded from the study due to lack of sufficient resources to pay for translator and interpreter services.
* Minors will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
T1 relaxometry value of Region of Interest (ROI) in MRF scan for each tumor type | At end of scan (45 minuets after beginning study)
T2 relaxometry value of Region of Interest (ROI) in MRF scan for each tumor type | At end of scan (45 minuets after beginning study)
Prediction analysis of MRF scans | At 6 months
Prediction analysis of MRF scans | At 9 months
Prediction analysis of MRF scans | At 12 months

SECONDARY OUTCOMES:
Number of patients whose clinical diagnosis and quantitative imaging diagnosis match | At end of scan (45 minuets after beginning study)
In treated tumors, difference in T1 relaxation times between baseline and 6 months post surgery | 6 months post-operative
In treated tumors, difference in T2 relaxation times between baseline and 6 months post surgery | 6 months post-operative
In treated tumors, difference in T1 and T2 relaxation times between recurrent tumor and radiation necrosis | At end of scan (45 minuets after beginning study)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra A Badve, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States